CLINICAL TRIAL: NCT04703322
Title: A Phase 2, Multicenter, Two-Part, Open-Label Study of Pexidartinib in Adult Subjects With Tenosynovial Giant Cell Tumor in Japan
Brief Title: A Study of Pexidartinib in Tenosynovial Giant Cell Tumor in Japan
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Daiichi Sankyo Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Daiichi Sankyo (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PL3397-A-J304; jRCT2041200074 (Other: Japan Registry of Clinical Trials)
Record Dates: First submitted 2020-12-22; First posted 2021-01-11 (Actual); Results first posted 2025-03-03 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Tenosynovial Giant Cell Tumor
Keywords: Tenosynovial Giant Cell Tumor; TGCT; Giant Cell Tumor of Tendon Sheath; GCTTS; Pigmented Villonodular Synovitis; PVNS
MeSH Terms: conditions — Giant Cell Tumor of Tendon Sheath; Synovitis, Pigmented Villonodular | interventions — pexidartinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Pexidartinib (Experimental): Participants with TGCT who will receive oral pexidartinib 800 mg (400 mg twice daily [BID]).
  Interventions: Drug: Pexidartinib

INTERVENTIONS:
Drug: Pexidartinib — 400 mg twice daily for a total daily dose of 800 mg (each capsule contains 200 mg of pexidartinib for oral administration)
  Other Names: TURALIO™; PLX3397

SUMMARY:
This phase 2, multicenter, two-part, open-label, single-arm study will be conducted in Japan and will evaluate the safety, tolerability, pharmacokinetics (PK), and efficacy of pexidartinib in adult participants with symptomatic tenosynovial giant cell tumor (TGCT) associated with severe morbidity or functional limitation and not amenable to improvement with surgery.

DETAILED DESCRIPTION:
This study will consist of 2 parts. In Part 1, pexidartinib 800 mg/day (400 mg twice a day [BID]) will be administered on an empty stomach and tolerability and PK of pexidartinib will be evaluated to determine the initiation of Part 2. In Part 2, pexidartinib 800 mg/day (400 mg BID) will be administered on an empty stomach and efficacy, safety, and PK of pexidartinib will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥20 years
* A diagnosis of TGCT (i) that has been histologically confirmed by a pathologist1 and (ii) associated with severe morbidity or functional limitations and not amenable to improvement with surgery determined consensually by qualified personnel (eg, 2 surgeons or a multi-disciplinary tumor board).
* Measurable disease as defined by RECIST version 1.1 (except that a minimal size of 2 cm is required), assessed from MRI scan by a central radiologist.

Exclusion Criteria:

* Known metastatic TGCT.
* Pre-existing increased serum transaminases; total bilirubin or direct bilirubin (>upper limit of normal); or active liver or biliary tract disease, including increased alkaline phosphatase.
* Significant concomitant arthropathy in the affected joint, serious illness, uncontrolled infection, or a medical or psychiatric history that, in the Investigator's opinion, would likely interfere with a participant's study participation or the interpretation of his or her results.
* Use of strong cytochrome P450 3A inducers, including St John's wort, proton pump inhibitors and potassium-competitive acid blockers, or other products known to cause hepatotoxicity.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2023-03-20 (Actual); Study Completion 2026-05-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (6):
- Japan (6):
  - Nagoya University Hospital, Aichi
  - Kyushu University Hospital, Fukuoka
  - Kanazawa University Hospital, Ishikawa
  - National Hospital Organization Osaka National Hospital, Osaka
  - Osaka International Cancer Institute, Osaka
  - National Cancer Center Hospital, Tokyo

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 9 participants who met all inclusion criteria and no exclusion criteria were enrolled in the study. These results are based on Part 1 of the study. All safety and pharmacokinetic primary outcome analysis data for Part 1 are reported. Part 2 of the study was not conducted. Eight patients remain in the study and are being followed until study completion. Only the final safety data of the patients who remain on study will be reported at the final database cut (estimated May 31, 2026).
Groups:
- Pexidartinib: Participants with TGCT who received oral pexidartinib 800 mg (400 mg twice daily [BID]).
Period: Overall Study
Arm/Group | Pexidartinib
Started | 9
Completed | 0
Not Completed | 9
Not completed — Ongoing | 8
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Demographic and baseline characteristics were assessed in the Safety Analysis Set.
Arm/Group | Pexidartinib
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.9 (11.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 9
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Dose-limiting Toxicity (DLT) in Part 1
Description: The number of participants with any-grade DLT treatment-emergent adverse events (TEAEs) were assessed.
Time Frame: Cycle 1, Day 1 to Cycle 1, Day 28 (each cycle is 28 days)
Population: All DLT TEAEs were assessed in the DLT Evaluable Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Pexidartinib
Number analyzed (Participants) | 9
Participants
  Any Grade DLT TEAE | 2
  Any Grade Hepatic function abnormal | 1
  Any Grade Alanine aminotransferase increased | 1
  Any Grade Aspartate aminotransferase increased | 1
  Any Grade Blood alkaline phosphatase increased | 1
  Any Grade Gamma-glutamyltransferase increased | 1

2. Primary Outcome: Pharmacokinetic Parameter Maximum Concentration of Pexidartinib and ZAAD-1006a (Cmax) in Part 1
Description: Pharmacokinetic parameters were assessed using non-compartmental methods. Cmax is the maximum concentration of pexidartinib and ZAAD-1006a in plasma.
Time Frame: Predose, 0.5 hours (hr), 1 hr, 2 hr, 4 hr, 6 hr, 8 hr, 24 hr post-dose of Cycle 1, Day 1 (C1D1) and Predose, 0.5 hr, 1 hr, 2 hr, 4 hr, and 6 hr postdose of Cycle 1, Day 15 (C1D15) (each cycle is 28 days)
Population: Pharmacokinetic data were assessed in the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Pexidartinib
Number analyzed (Participants) | 9
ng/mL
  Pexidartinib, C1D1 | 7920 (1720)
  Pexidartinib, C1D15: number analyzed (Participants) | 3
  Pexidartinib, C1D15 | 8810 (1110)
  ZAAD-1006a, C1D1 | 8000 (1990)
  ZAAD-1006a, C1D15: number analyzed (Participants) | 3
  ZAAD-1006a, C1D15 | 11700 (3340)

3. Primary Outcome: Pharmacokinetic Parameter Area Under the Concentration-Time Curve From Time Zero to Time of Last Measurable Concentration of Pexidartinib and ZAAD-1006a (AUClast) in Part 1
Description: Pharmacokinetic parameters were assessed using non-compartmental methods. AUClast is the area under the concentration-time curve from time zero to time of last measurable concentration of pexidartinib and ZAAD-1006a in plasma.
Time Frame: Predose, 0.5 hours (hr), 1 hr, 2 hr, 4 hr, 6 hr, 8 hr, 24 hrs post-dose of Cycle 1, Day 1 (C1D1) (each cycle is 28 days)
Population: Pharmacokinetic data were assessed in the Pharmacokinetic Analysis Set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Pexidartinib
Number analyzed (Participants) | 9
h*ng/mL
  Pexidartinib, C1D1 | 62000 (27.3)
  ZAAD-1006a, C1D1 | 90900 (48.4)

4. Primary Outcome: Pharmacokinetic Parameter Area Under the Concentration-Time Curve Up to Infinity of Pexidartinib and ZAAD-1006a (AUCinf) in Part 1
Description: Pharmacokinetic parameters were assessed using non-compartmental methods. AUCinf is the area under the concentration-time curve up to infinity of pexidartinib and ZAAD-1006a in plasma.
Time Frame: as for outcome 3
Population: Pharmacokinetic data were assessed in participants with available data in the Pharmacokinetic Analysis Set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Pexidartinib
Number analyzed (Participants) | 9
h*ng/mL
  Pexidartinib, C1D1 | 8700 (28.1)
  ZAAD-1006a, C1D1: number analyzed (Participants) | 7
  ZAAD-1006a, C1D1 | 195000 (40.2)

5. Primary Outcome: Pharmacokinetic Parameter Time to Reach Maximum Concentration of Pexidartinib and ZAAD-1006a (Tmax) in Part 1
Description: Pharmacokinetic parameters were assessed using non-compartmental methods. Tmax is the time to reach maximum concentration of pexidartinib and ZAAD-1006a in plasma.
Time Frame: as for outcome 2
Population: Pharmacokinetic data were assessed in the Pharmacokinetic Analysis Set.
Measure: Median (Full Range); unit: hours
Arm/Group | Pexidartinib
Number analyzed (Participants) | 9
hours
  Pexidartinib, C1D1 | 2.05 [1.97 to 2.10]
  Pexidartinib, C1D15: number analyzed (Participants) | 3
  Pexidartinib, C1D15 | 2.10 [1.92 to 2.15]
  ZAAD-1006a, C1D1 | 3.97 [1.97 to 7.92]
  ZAAD-1006a, C1D15: number analyzed (Participants) | 3
  ZAAD-1006a, C1D15 | 3.83 [2.10 to 3.92]

6. Primary Outcome: Objective Response Rate (ORR) Based on Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST Version 1.1) in Part 2
Description: ORR will be assessed by centrally reviewed MRI scan based on RECIST version 1.1. Complete response (CR) was defined as a disappearance of all target lesions, partial response (PR) was defined as at least a 30% decrease in the sum of diameters of target lesions, and stable disease (SD) was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD; at least a 20% increase in the sum of diameters of target lesions.
Time Frame: Week 25
Population: Part 2 of this study was not conducted and efficacy data are not available for reporting. Only the final safety data of patients who remain in the study will be reported at the final database cut (estimated May 31, 2026).
Arm/Group | Pexidartinib
Number analyzed (Participants) | 0

7. Secondary Outcome: ORR Based on Tumor Volume Score (TVS) in Part 2
Description: ORR will be assessed by centrally reviewed MRI scan based on TVS.
Time Frame: Week 25
Population: as for outcome 6
Arm/Group | Pexidartinib
Number analyzed (Participants) | 0

8. Secondary Outcome: Range of Motion (ROM) in Part 2
Description: Mean change from baseline in ROM of the affected joint, relative to a reference standard for the same joint will be assessed.
Time Frame: Week 25
Population: as for outcome 6
Arm/Group | Pexidartinib
Number analyzed (Participants) | 0

9. Secondary Outcome: Patient-reported Outcomes Measurement Information System (PROMIS) Physical Function Scale in Part 2
Description: Mean change from baseline score in the PROMIS Physical Function Scale will be assessed.
Time Frame: Week 25
Population: as for outcome 6
Arm/Group | Pexidartinib
Number analyzed (Participants) | 0

10. Secondary Outcome: Brief Pain Inventory (BPI) Worst Pain Numeric Rating Scale (NRS) in Part 2
Description: Proportion of responders will be assessed based on the BPI Worst Pain NRS item and analgesic use by BPI-30 definition (ie, 30% or more improvement in average NRS).
Time Frame: Week 25
Population: as for outcome 6
Arm/Group | Pexidartinib
Number analyzed (Participants) | 0

11. Secondary Outcome: Best Overall Response (BOR) Based on RECIST Version 1.1 in Part 2
Description: BOR will be assessed by centrally reviewed magnetic resonance imaging (MRI) scan based on RECIST version 1.1.
Time Frame: Post Week 25 visit or following discontinuation from Part 2 of the study (whichever occurs first), up to approximately 1 year 6 months
Population: as for outcome 6
Arm/Group | Pexidartinib
Number analyzed (Participants) | 0

12. Secondary Outcome: BOR Based on TVS in Part 2
Description: BOR will be assessed by centrally reviewed MRI scan based on TVS.
Time Frame: as for outcome 11
Population: as for outcome 6
Arm/Group | Pexidartinib
Number analyzed (Participants) | 0

13. Secondary Outcome: Duration of Response (DoR) Based on RECIST Version 1.1 in Part 2
Description: DoR will be assessed by centrally reviewed MRI scan based on RECIST version 1.1.
Time Frame: as for outcome 11
Population: as for outcome 6
Arm/Group | Pexidartinib
Number analyzed (Participants) | 0

14. Secondary Outcome: DoR Based on TVS
Description: DoR will be assessed by centrally reviewed MRI scan based on TVS.
Time Frame: as for outcome 11
Population: as for outcome 6
Arm/Group | Pexidartinib
Number analyzed (Participants) | 0

15. Secondary Outcome: Number of Participants Reporting Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events
Time Frame: Baseline up to 28 (+/- 7 days) after last dose, up to approximately 6 years 9 months
Reporting Status: Not Posted, anticipated posting 2027-05

ADVERSE EVENTS:
Time Frame: Adverse events were collected from screening to 28 days (+/-7 days) after last dose of study treatment, up to 3 years 7 months (data cut-off date).
Arm/Group | Pexidartinib
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 9/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pexidartinib (N=9)
Hair colour changes (Skin and subcutaneous tissue disorders) | 7
Pruritus (Skin and subcutaneous tissue disorders) | 4
Dermatitis (Skin and subcutaneous tissue disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 1
Skin discolouration (Skin and subcutaneous tissue disorders) | 1
Aspartate aminotransferase increased (Investigations) | 7
Alanine aminotransferase increased (Investigations) | 4
Blood lactate dehydrogenase increased (Investigations) | 3
Gamma-glutamyltransferase increased (Investigations) | 3
Blood alkaline phosphatase increased (Investigations) | 2
Blood bilirubin increased (Investigations) | 2
Blood creatinine phosphokinase increased (Investigations) | 2
Blood creatinine increased (Investigations) | 2
Neutrophil count decreased (Investigations) | 2
Amylase increased (Investigations) | 1
Blood cholesterol increased (Investigations) | 1
Weight decreased (Investigations) | 1
Pyrexia (General disorders) | 2
Face oedema (General disorders) | 1
Fatigue (General disorders) | 1
COVID-19 (Infections and infestations) | 2
Norovirus infection (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Anaemia (Blood and lymphatic system disorders) | 1
Eosinophilia (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 2
Dysgeusia (Nervous system disorders) | 2
Hypertension (Vascular disorders) | 2
Hypokalaemia (Metabolism and nutrition disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-08-27): https://cdn.clinicaltrials.gov/large-docs/22/NCT04703322/Prot_SAP_000.pdf